CLINICAL TRIAL: NCT03106493
Title: Upstate New York Infant Development Screening Program
Acronym: Upstate KIDS
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: New York State Department of Health (Other Government); University at Albany (Other)
Responsible Party: Sponsor
Other Study IDs: HHSN275201400013C
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Obesity; Blood Pressure; Motor Delay; Developmental Delay; Asthma; Allergies
MeSH Terms: conditions — Obesity; Psychomotor Disorders; Learning Disabilities; Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, urine, saliva (in subgroup under ongoing future work)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary: Singletons and 1 twin of each pair
  Interventions: Other: None (observational)
- Secondary: Twin sibling of children enrolled in primary cohort
  Interventions: Other: None (observational)
- Tertiary: Higher order multiples and siblings
  Interventions: Other: None (observational)

INTERVENTIONS:
Other: None (observational) — None (observational)

SUMMARY:
The goal of the Upstate KIDS Study is to track the growth, development and long-term health of children given the increasing use of infertility treatment, occurrence of maternal obesity and pregnancy complications, and rising maternal age at birth.

DETAILED DESCRIPTION:
The Upstate KIDS Study aims to determine if there are differences in health measures between children conceived by infertility treatment and children conceived naturally. In the first phase of the study, the focus was on growth and development through age 3 years. In the second phase of the study, the focus is turning to cardiometabolic factors through age 9 years. Infertility treatments include assisted reproductive technologies (ART) such as in vitro fertilization (IVF), controlled ovarian hyperstimulation (COH) and ovulation induction (OI). The study was originally designed as a matched exposure cohort. Specifically, singletons whose birth certificates indicated the use of infertility treatment were considered 'exposed' singleton infants and subsequently frequency-matched on perinatal region of birth at a ratio of 1:3 to 'unexposed' singletons. Twins and higher order multiples were invited to participate regardless of mode of conception. Mothers and their newborns were recruited approximately 2-4 months postpartum. The first phase of the study was completed in 2014 and main findings can be found under publications.

The second phase objectives are:

To determine whether infertility treatment is associated with differences in growth and development from age 6 to 8 years with particular focus on childhood cardio-metabolic outcomes by follow-up of children conceived by ART or other infertility treatments and children who were conceived without treatment. Secondarily, to assess epigenetic differences as measured by DNA methylation using collected biospecimens.

ELIGIBILITY:
Inclusion Criteria:

* Mothers delivering a live birth in New York State (excluding New York City).

Exclusion Criteria:

* Refused follow-up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Exposure enriched cohort as described: Buck Louis GM, Hediger ML, Bell EM, Kus CA, Sundaram R, McLain AC, Yeung E, Hills EA, Thoma ME, Druschel CM. Methodology for Establishing a Population-Based Birth Cohort Focusing on Couple Fertility and Children's Development, the Upstate KIDS Study. Paediatric and Perinatal Epidemiology. 2014 May;28(3):191-202.
Sampling Method: Non-Probability Sample
Enrollment: 6171 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Through age 9 years
  Measurement of blood pressure

SECONDARY OUTCOMES:
Motor milestone development | 4-24 months
  Study collected information using questionnaires to mothers with aid of journal

OTHER OUTCOMES:
Breastfeeding information | 4-12 months
  Study collected information using questionnaires to mothers

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available for public use by NIH data sharing system.

REFERENCES:
- [Background] Buck Louis GM, Hediger ML, Bell EM, Kus CA, Sundaram R, McLain AC, Yeung E, Hills EA, Thoma ME, Druschel CM. Methodology for establishing a population-based birth cohort focusing on couple fertility and children's development, the Upstate KIDS Study. Paediatr Perinat Epidemiol. 2014 May;28(3):191-202. doi: 10.1111/ppe.12121. Epub 2014 Mar 25. PMID 24665916
- [Background] Andersen NJ, Mondal TK, Preissler MT, Freed BM, Stockinger S, Bell E, Druschel C, Louis GM, Lawrence DA. Detection of immunoglobulin isotypes from dried blood spots. J Immunol Methods. 2014 Feb;404:24-32. doi: 10.1016/j.jim.2013.12.001. Epub 2013 Dec 13. PMID 24333851
- [Background] Buck Louis GM, Druschel C, Bell E, Stern JE, Luke B, McLain A, Sundaram R, Yeung E. Use of assisted reproductive technology treatment as reported by mothers in comparison with registry data: the Upstate KIDS Study. Fertil Steril. 2015 Jun;103(6):1461-8. doi: 10.1016/j.fertnstert.2015.02.033. Epub 2015 Mar 23. PMID 25813287
- [Background] Yeung EH, Sundaram R, Bell EM, Druschel C, Kus C, Ghassabian A, Bello S, Xie Y, Buck Louis GM. Examining Infertility Treatment and Early Childhood Development in the Upstate KIDS Study. JAMA Pediatr. 2016 Mar;170(3):251-8. doi: 10.1001/jamapediatrics.2015.4164. PMID 26746435
- [Background] Yeung EH, Sundaram R, Bell EM, Druschel C, Kus C, Xie Y, Buck Louis GM. Infertility treatment and children's longitudinal growth between birth and 3 years of age. Hum Reprod. 2016 Jul;31(7):1621-8. doi: 10.1093/humrep/dew106. Epub 2016 May 10. PMID 27165624
- [Derived] Clayton PK, Putnick DL, Trees IR, Robinson SL, O'Connor TG, Tyris JN, Yeung EH. Age of Juice Introduction and Cardiometabolic Outcomes in Middle Childhood. J Nutr. 2024 Aug;154(8):2514-2523. doi: 10.1016/j.tjnut.2024.06.014. Epub 2024 Jun 26. PMID 38936550
- [Derived] Polinski KJ, Robinson SL, Putnick DL, Sundaram R, Ghassabian A, Joseph P, Gomez-Lobo V, Bell EM, Yeung EH. Maternal self-reported polycystic ovary syndrome with offspring and maternal cardiometabolic outcomes. Hum Reprod. 2024 Jan 5;39(1):232-239. doi: 10.1093/humrep/dead227. PMID 37935839
- [Derived] Yeung EH, Mendola P, Sundaram R, Lin TC, Broadney MM, Putnick DL, Robinson SL, Polinski KJ, Wactawski-Wende J, Ghassabian A, O'Connor TG, Gore-Langton RE, Stern JE, Bell E. Conception by fertility treatment and cardiometabolic risk in middle childhood. Fertil Steril. 2022 Aug;118(2):349-359. doi: 10.1016/j.fertnstert.2022.04.030. Epub 2022 Jun 10. PMID 35697532
- [Derived] Michels KA, Ghassabian A, Mumford SL, Sundaram R, Bell EM, Bello SC, Yeung EH. Breastfeeding and motor development in term and preterm infants in a longitudinal US cohort. Am J Clin Nutr. 2017 Dec;106(6):1456-1462. doi: 10.3945/ajcn.116.144279. Epub 2017 Nov 1. PMID 29092884